CLINICAL TRIAL: NCT03468153
Title: The Safety and Efficacy of Dual Specificity CD19 and CD22 CAR-T Cell Immunotherapy for CD19+CD22+ Relapsed and Refractory Lymphoma
Brief Title: Dual Specificity CD19 and CD22 CAR-T Cell Immunotherapy for CD19+CD22+ Relapsed and Refractory Lymphoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Collaborators: Shanghai Unicar-Therapy Bio-medicine Technology Co.,Ltd (Industry)
Responsible Party: Principal Investigator, Zhao Weili, Professor, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ruijin-CAR-01
Record Dates: First submitted 2018-03-11; First posted 2018-03-16 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T cell therapy (Experimental): Patient-derived dual specificity CD19 and CD22 CAR-T
  Interventions: Biological: Dual Specificity CD19 and CD22 CAR-T Cell Immunotherapy

INTERVENTIONS:
Biological: Dual Specificity CD19 and CD22 CAR-T Cell Immunotherapy — Patient-derived dual specificity CD19 and CD22 CAR-T Cells

SUMMARY:
Patients with relapsed or refractory lymphoma often develop resistance to chemotherapy. Chimeric antigen receptor-modified T cell (CART) therapy showed promising effect in B-cell malignancies these years. CD19 and CD22 are proteins expressed on the surface of the lymphoma cells in patients with CD19+CD22+ lymphoma. The CAR enables the T-cells to recognize and kill the tumor cell through recognition of CD19 and CD22. This is a phase 2 trial to study the safety and efficacy of dual specificity CD19 and CD22 CAR-T cell immunotherapy for CD19+CD22+ relapsed and refractory lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Histological detection confirmed CD19/CD22 postive lymphoma;
* Recieved more than 2 lines of chemotherapy;
* Not eligible for hematopoietic stem cell transplantation or relapsed after hematopoietic stem cell transplantation;
* Life expectation for more than 3 months;
* ECOG ≥ 2;
* Adequate organ function: EF≥50%; normal ECG; CCR≥40ml/min; ALT and AST ≤ 3 × upper limitation of normal, T-BIL ≤ 2.0mg/dl; PT and APTT < 2 × upper limitation of normal; SpO2 > 92%;
* CBC results: Hb ≥ 80g/L, ANC > 1 × 10E9/L, Plt ≥ 50 × 10E9/L;
* Results of pregnant test should be negative, and agree to conception control during treatment and 1 year after CAR-T infusion;
* With measurable disease;
* Written informed consent could be acquired;

Exclusion Criteria:

* Immunosuppressive agents or steroids in recent 1 week before recruitment;
* Uncontrolled infection;
* HIV positive ;
* Active HBV or HCV infection;
* Women in pregnancy and lactation;
* Refuse to conception control during treatment and 1 year after CAR-T infusion;
* Uncured malignancies other than non-Hodgkin lymphoma;
* Have participated similar trial for treating relapse/refractory non-Hodgkin lymphoma;
* Inheritated immune deficiancy;
* Severe heart disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Overall remission rate | 4 weeks after infusion
  Rate of complete remission and patial remission

SECONDARY OUTCOMES:
Adverse toxicity | Day 0, day 4, week 1, week 3, week 4, month 2, month 12 after CAR-T cells were infused
  According to CTCAE 4.0 criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided